CLINICAL TRIAL: NCT06332950
Title: A Randomized, Multi-cohort, Multi-center Phase Ib/II Study of Adebrelimab Plus Irinotecan Liposome (II) With or Without Famitinib in Patients With ES-SCLC Pre-treated With Immune Checkpoint Inhibitor(s)
Brief Title: Safety and Efficacy of Adebrelimab Plus Irinotecan Liposome (II) With or Without Famitinib in ES-SCLC Pre-treated With Immunotherapy
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baohui Han (Other)
Responsible Party: Sponsor-Investigator, Baohui Han, Chief physician, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-SCLC-II-015
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — irinotecan sucrosofate; famitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adebrelimab plus Irinotecan Liposome (II) (Experimental): Adebrelimab: 1200 mg, IV, D1, Q3W
  Irinotecan Liposome (II): RP2D, IV, D1, Q3W
  Interventions: Drug: Adebrelimab, Irinotecan Liposome (II)
- Adebrelimab plus Irinotecan Liposome (II) and Famitinib (Experimental): Adebrelimab: 1200 mg, IV, D1, Q3W
  Irinotecan Liposome (II): RP2D, IV, D1, Q3W
  Famitinib: RP2D, QO, QD
  Interventions: Drug: Adebrelimab, Irinotecan Liposome (II), Famitinib

INTERVENTIONS:
Drug: Adebrelimab, Irinotecan Liposome (II) — Adebrelimab:1200 mg, IV, D1, Q3W
  Irinotecan Liposome (II): RP2D, IV, D1, Q3W
  Escalating doses to determine recommended phase 2 dose (RP2D) of Irinotecan Liposome (II).
  Participants will receive Adebrelimab (1200 mg, IV, D1, Q3W) plus the RP2D of Irinotecan Liposome (II).
  Arms: Adebrelimab plus Irinotecan Liposome (II)
Drug: Adebrelimab, Irinotecan Liposome (II), Famitinib — Adebrelimab:1200 mg, IV, D1, Q3W
  Irinotecan Liposome (II): RP2D, IV, D1, Q3W
  Famitinib: RP2D, QO, QD
  Escalating doses to determine recommended phase 2 dose (RP2D) of Famitinib.
  Participants will receive Adebrelimab (1200 mg, IV, D1, Q3W) plus the RP2D of Irinotecan Liposome (II) and Famitinib.
  Arms: Adebrelimab plus Irinotecan Liposome (II) and Famitinib

SUMMARY:
This is an open-label, randomized, multi-cohort, multi-center, phase Ib/II study to evaluate the safety and efficacy of Adebrelimab plus Irinotecan Liposome (II) with or without Famitinib in patients with extensive-stage small cell lung cancer (ES-SCLC) pre-treated with immune checkpoint inhibitor(s).

DETAILED DESCRIPTION:
This study is divided into two stages. Dose exploration will be conducted first, and after obtaining preliminary safety data it will be decided by investigator when to proceed with dose extension. The aim of this study is to observe and evaluate the safety and efficacy of Adebrelimab plus Irinotecan Liposome (II) with or without Famitinib.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate and sign the informed consent form.
* Age: 18-75 years old, male or female.
* ECOG PS: 0-1 points.
* Histologically or cytologically confirmed of extensive stage small cell lung cancer (according to the International Association for the Study of Lung Cancer, 8th Edition or VALG II staging system).
* Progression after first-line immunotherapy combined with platinum-based system therapy more than 90 days.
* At least one measurable lesion (RECIST 1.1 criteria) was assessed by imaging evaluation (enhanced CT or MRI) within 4 weeks prior to enrollment.
* Patients with asymptomatic or treatment-stabilized central nervous system (CNS) metastases must meet the following conditions: (1) No imaging progress for at least 4 weeks after the end of treatment; (2) completion of treatment 4 weeks before enrollment; (3) no treatment with systemic corticosteroids (>10mg/ day prednisone or other equivalent dose) within the first 2 weeks before enrollment.
* Expected survival time ≥12 weeks.
* Adequate hematology and organ function (No blood transfusion or blood products, no correction with G-CSF and other hematopoietic stimulating factors within 14 days), including:

  1. Complete blood count: White blood cell count WBC≥3.0×109/L; Absolute neutrophil count ANC≥1.5×109/ L; Platelet count≥100×109/ L; Hemoglobin≥90 g/L.
  2. Liver function: AST≤2.5× upper limit of normal(ULN); ALT≤2.5×ULN (Patients with liver metastasis, AST and ALT≤5×ULN); TBIL≤1.5×ULN (Except for Gilbert syndrome ≤3×ULN); ALB≥30.0 g/L.
  3. Renal function: Serum creatinine≤1.5×ULN or creatinine clearance≥50ml/min (Cockcroft-Gault formula).
  4. Normal coagulation function: INR and APTT≤1.5×ULN.
  5. TSH≤ULN.
  6. Other: Lipase≤1.5×ULN (Patients with lipase>1.5×ULN but no clinical or imaging evidence of pancreatitis could be enrolled); Amylase≤1.5×ULN (Patients with amylase >1.5×ULN but no clinical or imaging evidence of pancreatitis could be enrolled); ALP≤2.5×ULN (Patients with bone metastasis, ALP≤5×ULN).
  7. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF)≥50%.
* Women of childbearing potential must undergo a negative pregnancy test (HCG) 7 days prior to initiation of treatment, and women of childbearing potential and men (who are sexually active with women of childbearing potential) must agree to use effective contraception uninterruptedly for the duration of the treatment period and for 3 months after the administration of the last therapeutic dose.

Exclusion Criteria:

* Non-small cell lung cancer or non-small cell lung cancer admixed with components of small cell lung cancer, as confirmed by histology or cytology.
* With > 2 lines of prior chemotherapy.
* Patients previously treated with topoisomerase I inhibitors.
* With primary resistance, defined as patients who do not respond to first-line treatment or progress within 90 days after the end of treatment.
* Patients previously treated with antiangiogenic drugs, such as bevacizumab, recombinant human endostatin, anlotinib, apatinib, etc.
* Radiotherapy for the chest and whole brain was completed within 4 weeks prior to enrollment (enrollment was allowed if palliative radiotherapy for bone lesions could complete before the first dose).
* Except for alopecia and fatigue, toxicity due to previous antitumor therapy did not recover to CTCAE 5.0≤1 level before enrollment. Other toxicities due to previous antitumor therapy are not expected to resolve and have long-lasting sequelae.
* With active brain metastasis or meningeal metastasis. Compressive myelopathy that has not been cured or alleviated after surgery and/or radiotherapy, or present with compressive paraplegia or paraplegia after treatment in patients previously diagnosed with compressive myelopathy. Patients with liver metastases had significant clinical symptoms and abnormal liver function after cryotherapy and radiofrequency ablation treatment within the first 4 weeks of enrollment. Patients with uncontrolled mass pleural effusion, pericardial effusion, or ascites. Patients with cardiovascular disease.
* Patients previously treated with systemic immunosuppressive medications within 4 weeks before enrollment.
* Presence or history of active autoimmune disease. Interstitial pneumonia, drug-induced pneumonia, radiation pneumonia requiring steroid treatment (greater than 10 mg/day prednisone or its equivalent), or active pneumonia with clinical symptoms.
* Patients with an active or uncontrolled severe infection (CTCAE 5.0≥2) within 2 weeks prior to the first dose.
* With active tuberculosis or tuberculosis under treatment.
* Congenital or acquired immunodeficiency, such as human immunodeficiency virus (HIV) infection. Untreated active hepatitis B (HBsAg positive or HBV DNA≥500 IU/ml with abnormal liver function), hepatitis C (hepatitis C antibody positive, with higher HCV-RNA than the lower detection limit of the assay method and abnormal liver function) or hepatitis B and C co-infection.
* Hypertension that cannot be controlled with medications (systolic blood pressure≥140 mmHg or diastolic blood pressure≥90 mmHg). History of hypertensive crisis or hypertensive encephalopathy.
* Arteriovenous thrombosis events occurred within 24 weeks prior to signing the ICF, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism.
* With factors influencing absorption of drug, such as refractory nausea and vomiting, chronic gastrointestinal diseases, or inability to swallow the formulated product.
* With mental illness, alcoholism, inability to quit smoking, drug or substance abuse.
* With known allergic history of the drug components of this program, or allergic to other monoclonal antibodies.
* Received any other investigational treatment or participated in any other interventional clinical trials within 4 weeks prior to signing the ICF.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival | Up to 6 months
  Proportion of disease progression or death from randomization to 6 months of treatment.

SECONDARY OUTCOMES:
Safety | Up to 3 months after the last dose
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.
Objective response rate | Up to 36 months
  Objective response rate, determined according to RECIST v1.1 criteria.
Progression-free survival | Up to 36 months
  Progression Free Survival, determined according to RECIST v1.1 criteria.
Overall survival | Up to 36 months
  Overall survival is the time from randomization to death due to any reason or loss of follow-up.
Disease control rate | Up to 36 months
  Disease Control Rate, determined according to RECIST v1.1 criteria.
Duration of response | Up to 36 months
  Duration of Response, determined according to RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No